CLINICAL TRIAL: NCT00003860
Title: Intensive Chemotherapy With Peripheral Blood Stem Cell Support for Small Cell Lung Cancer
Brief Title: Combination Chemotherapy Plus Peripheral Stem Cell Transplantation in Treating Patients With Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067023; FRE-FNCLCC-98003-CLEO; EU-98072; FRE-FNCLCC-CLEOPATRE03
Record Dates: First submitted 1999-11-01; First posted 2004-06-16 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Filgrastim; Carboplatin; Etoposide; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: etoposide
Drug: ifosfamide
Procedure: in vitro-treated peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus peripheral stem cell transplantation in treating patients who have small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility of the administration of intensive chemotherapy with ifosfamide, carboplatin, and etoposide followed by peripheral blood stem cell support in patients with small cell lung cancer. II. Determine the rate and duration of response in these patients after this treatment. III. Determine the progression free and overall survival of these patients.

OUTLINE: This is an open label, multicenter study. Patients receive 4 courses of intensive chemotherapy consisting of ifosfamide IV over 24 hours and carboplatin IV over 1 hour on day 1 and etoposide IV over 1 hour on days 1 and 2. Filgrastim (G-CSF) is administered subcutaneously beginning on day 2 and continuing until blood cell counts recover. Courses repeat every 14 days. Peripheral blood stem cells (PBSC) are collected after course 1. PBSC are reinfused on day 3 of courses 2 and 3. Patients who experience a complete response receive prophylactic cerebral irradiation on day 71. Patients are followed every 2 months for 5 years.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven small cell lung cancer Good prognosis on the Manchester scale, with no more than 2 of the following high risk factors: Karnofsky less than 60% Hyponatremia (low sodium) Alkaline phosphatase at least 1.5 times upper limit of normal (ULN) LDH greater than ULN No symptomatic CNS metastases requiring corticosteroids

PATIENT CHARACTERISTICS: Age: 18 to 60 Performance status: See Disease Characteristics Life expectancy: Not specified Hematopoietic: Neutrophil count at least 2,000/mm3 Platelet count at least 125,000/mm3 Hepatic: See Disease Characteristics Bilirubin less than 1.25 times upper limit of normal (ULN) SGOT/SGPT less than 1.25 times ULN Renal: Creatinine less than ULN Cardiovascular: LVEF at least 50% No myocardial infarction within 5 years No uncontrolled cardiac disease Pulmonary: No severe chronic obstructive pulmonary disease Other: No neurological symptoms greater than grade 2 No severe psychoses No other concurrent medical problems No active infection HIV negative No allergy to E. coli derived products No prior malignancy within 5 years except basal cell skin cancer, carcinoma in situ of the cervix, or lung or respiratory cancer in remission Not pregnant or nursing

PRIOR CONCURRENT THERAPY: See Disease Characteristics No prior antineoplastic therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 1998-09 (Actual); Primary Completion 2000-08 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronique N. Trillet-Lenoir, MD, Study Chair — Centre Hospitalier Lyon Sud
Locations (22):
- France (22):
  - CHR de Besancon - Hopital Saint-Jacques, Besançon
  - Institut Bergonie, Bordeaux
  - CMC Bligny, Briis-sous-Forges
  - Centre de Lute Contre le Cancer,Georges-Francois Leclerc, Dijon
  - CHR de Grenoble - La Tronche, Grenoble
  - Centre Leon Berard, Lyon
  - Hopital Louis Pradel, Lyon
  - Institut J. Paoli and I. Calmettes, Marseille
  - Hopital Arnaud de Villeneuve, Montpellier
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Institut Curie - Section Medicale, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Tenon, Paris
  - Hopital Jules Courmont - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hopital Rene Dubos, Pontoise
  - Institut Jean Godinot, Reims
  - Centre Rene Huguenin, Saint-Cloud
  - Hopitaux Universitaire de Strasbourg, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - CHRU de Nancy - Hopitaux de Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif